CLINICAL TRIAL: NCT03785730
Title: Impact of Non-restorative Cavity Control on Proximal Carious Lesions of Anterior Primary Teeth on the Tooth Survival and Patient-centered Outcomes (CEPECO 2) - Study Protocol for a Non-inferiority Randomized Clinical Trial
Brief Title: Non-restorative Cavity Control in Anterior Cavitated Caries Lesion of Primary Teeth
Acronym: CEPECO2
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Outbreak of COVID-19.
Sponsor: Universidade Ibirapuera (Other)
Responsible Party: Principal Investigator, Tamara Kerber Tedesco, Principal investigator, Universidade Ibirapuera
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unib3
Record Dates: First submitted 2018-12-18; First posted 2018-12-24 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-restorative cavity control - NRCC (Experimental): Enlargement with metallic sandpaper associated with toothbrushing/1000 ppm fluoride toothpaste.
  Interventions: Procedure: Non-restorative cavity control - NRCC group
- Resin composite restoration - RCR (Active Comparator): Selective carious lesion removal and restoration with resin composite.
  Interventions: Procedure: Restoration with resin composite - RCR group

INTERVENTIONS:
Procedure: Non-restorative cavity control - NRCC group — The proximal cavities will be enlarged with metallic sandpaper, exposing the cavity, to allow access for toothbrushing associated with 1000 ppm fluoride toothpaste.
  Arms: Non-restorative cavity control - NRCC
Procedure: Restoration with resin composite - RCR group — In control group, the treatment will be performed after prophylaxis and relative isolation. The selective carious tissue removal will be performed with appropriate dentin curettes. The acid conditioning will be performed only in enamel for 15 s with 37% phosphoric acid gel, and then the application of the adhesive system and restoration of resin composite will be conducted.
  Arms: Resin composite restoration - RCR

SUMMARY:
Background: Studies have questioned the necessity of restoring cavitated carious lesion on primary teeth, once the control of biofilm is the most important factor to arrest these lesions. This randomized clinical trial aimed to compare the survival of teeth treated with a non-restorative cavity control (NRCC) compared to resin composite restorations (RCR) on proximal carious lesion in anterior primary teeth, as well as the impact of these treatments on patient-centered outcomes. Methods: A randomized clinical trial with two parallels arms (1:1) will be conducted. Children between 3 and 6 years old will be selected from the Center of Clinic Research of Pediatric Dentistry of Ibirapuera University (UNIB), a dental trailer (FOUSP) located on Educational Complex Professor Carlos Osmarinho de Lima, the Pediatric Dentistry Clinic of Santa Cecília University and from the Pediatric Dentistry Clinic of University Center UNINOVAFAPI. One hundred and forty-eight teeth will be randomly distributed in two experimental groups: (1) Selective removal of carious tissue and RCR; or (2) NRCC through cavity enlargement using metallic sandpaper. The primary outcome will be tooth survival after 6, 12, 18, and 24 months. The duration and the cost of dental treatments will be considered for the estimation of the cost-effectiveness of the evaluated treatments. The discomfort reported by the participants will be measured after each treatment using the FIS scale. The participants' satisfaction and perception of the parents/legal guardians will be evaluated through questionnaires. For the primary outcome, Kaplan-Meier's survival and Long-Rank test will be used for comparison between the two groups. All the variables will be modeled by Cox regression with shared fragility. Significance will be considered at 5%.

DETAILED DESCRIPTION:
This non-inferiority randomized controlled clinical trial, with two parallel groups with 1:1 allocation ratio, was approved by the Research Ethics Committee of Universidade Ibirapuera (UNIB). The other centers involved are considered co-participants (Centro Universitário do Norte - Uninorte , Centro Universitário Uninovafapi - UNINOVAFAPI, and School of Dentistry from the University of Sao Paulo - FOUSP). Children aged 3 to 6 years with at least one proximal cavitated lesion on anterior primary teeth will be selected from the Clinical Pediatric Research Center. Teeth will be randomly allocated to selective removal of carious tissue and resin composite restoration (RCR) or NRCC. Tooth survival after two years of follow-up will be the primary outcome and cost-effectiveness, satisfaction, and discomfort reported by participants and parents/guardians' perception will be the secondary outcomes. Only patients who fulfill the eligibility criteria will be included in the study after the legal guardians sign the informed consent form and the child consents to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included that have at least one anterior tooth with carious lesion cavitated affecting the proximal surface.

Exclusion Criteria:

* Patients will be excluded with special needs, using orthodontics devices and/or systemic diseases which may affect the oral cavity.
* Also, teeth with lesions affecting more than one third of the buccal/lingual surfaces, with previous history of dental trauma, presenting pulp exposure, spontaneous pain, pathological mobility, presence of abscess or fistula next to the tooth, teeth with restorations, developmental enamel defects or physiological mobility (exfoliation) will be excluded.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Tooth survival by clinical assessment | 24 months
  Comparing the survival of teeth treated with restoration of resin composite and with NRCC for lesions cavitated in anterior primary teeth by clinical assessment, considering as success when the teeth will be without clinical signs or symptoms of pulp pathology or exfoliated, with no need for more invasive interventions, such as pulpectomy or extraction.

SECONDARY OUTCOMES:
Discomfort regarding the treatment options by a Face image scale (FIS) | Immediately after treatment
  Children-reported discomfort regarding the treatment options by a Face image scale (FIS). The scale present 5 different faces since "very happy" (scored as 1) until "very sad" (scored as 5) with the treatment. Higher scores mean a worse discomfort.
Cost-effectiveness analysis | 24 months.
  The duration of the treatments (time of treatment) and the cost of the materials used will be considered for the estimation of the cost-efficacy of the treatments by a ratio - cost/effectiveness, being effectiveness considered the tooth survival.
Perception of parents / guardians evaluated through questionnaire | Prior to treatment, immediately after and 6 months later.
  Parents perception of the treatments will be evaluated through a questionnaire - "Child's and parent's questionnaire about teeth appearance" - with possible answers varying from very satisfied until insatisfied. After the questionnaire is applied for the parents/guardians, the anwsers will bem transformed in scores 1 to 5, in according the original paper that validated the questionnaire. Higher scores mean a worse perception.
Satisfaction of children: questionnaire | After 6 months
  Children-reported satisfaction regarding the treatment by a questionnaire with five question which for answers will be used a Face image scale (FIS). The scale present 5 different faces since "very happy" (scored as 1) until "very sad" (scored as 5) with the treatment. Lower scores mean a better satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Tamara Kerber Tedesco, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available on Mendeley database.

REFERENCES:
- [Derived] Bianchi RMD, Pascareli-Carlos AM, Floriano I, Raggio DP, Braga MM, Gimenez T, Holanda MC, da Silva GS, de Natal KH, Tedesco TK. Impact of non-restorative cavity control on proximal carious lesions of anterior primary teeth on the tooth survival and patient-centered outcomes (CEPECO 2): study protocol for a non-inferiority randomized clinical trial. BMC Oral Health. 2021 Mar 31;21(1):167. doi: 10.1186/s12903-021-01524-0. PMID 33789643